CLINICAL TRIAL: NCT02187770
Title: Precision of IMED-4 Lung Fluid Measurements
Status: Completed | Type: Observational
Sponsor: Intersection Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-000040
Record Dates: First submitted 2014-07-07; First posted 2014-07-11 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Dyspnea; Acute Heart Failure Syndrome; Pulmonary Congestion
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: IMED-4 — Non invasive recording electrode used to assess lung fluid

SUMMARY:
The purpose of this study is to determine if IMED-4 recordings have sufficient precision to detect a clinically significant change in lung fluid status in acute heart failure syndrome with pulmonary congestion.

DETAILED DESCRIPTION:
The study will evaluate if the IMED-4 system has the precision to detect a clinically significant change in lung fluid status for patients with confirmed acute heart failure syndrome with pulmonary congestion. Changes in lung fluid in acute heart failure syndrome are difficult to diagnose and evaluate.

ELIGIBILITY:
Inclusion Criteria

1. Diagnosed with acute heart failure syndrome with pulmonary congestion defined by a Brain natriuretic peptide (BNP) >350 pg/mL or N-terminal pro-brain natriuretic peptide (NT-pro BNP) >1500 pg/mL and any one of the following:

   1. PCWP >25mmHg
   2. Dyspnea at rest in a recumbent sitting position (30 to 45 degrees), which has worsened within the past week
   3. Radiological evidence of CHF on a chest X-ray
   4. Physical exam as evidence for pulmonary congestion:

   i. Presence of an S3 heart sound ii. Lung rales/crackles/crepitations
2. Age greater than or equal to (≥) 18
3. Ability to reliably carry out self-assessment of symptoms
4. Willingness, ability and commitment to participate in index and follow-up IMED-4 recordings

EXCLUSION Criteria

1. Known active myocarditis, obstructive hypertrophic cardiomyopathy, constrictive pericarditis, uncorrected clinically significant primary valvular disease
2. Clinical diagnosis of acute coronary syndrome meeting any 2 of the following 3 criteria:

   1. Prolonged chest pain at rest, or an accelerated pattern of angina
   2. Electrocardiogram changes indicative of ischemia or myocardial injury
   3. Serum troponin >3 times upper limit of lab normal
3. Clinically-suspected acute mechanical cause of ADHF (e.g., papillary muscular rupture); the diagnosis need not be confirmed by imaging or cardiac catheterization
4. Estimated Glomerular Filtration Rate: eGFR <30mL/min/1.73m
5. Known vasculitis, active infective endocarditis, or suspected infections including pneumonia, acute hepatitis, systemic inflammatory response syndrome, or sepsis
6. Body temperature ≥38°C just prior to enrollment
7. Acute or chronic respiratory disorder (e.g. severe chronic obstructive pulmonary disease (COPD)) or primary pulmonary hypertension sufficient to cause dyspnea at rest, which may interfere with the ability to interpret dyspnea assessments or hemodynamic measurements
8. Total Albumin <2.5 g/dL
9. Patients requiring mechanical circulatory support
10. Pregnancy or lactation
11. Patients who have tattoos and/or non-intact skin directly under the electrode sensor position
12. Patients who have had past allergic reactions to medical grade adhesives
13. Patients who have had a lung lobectomy
14. Patients who decline to have their backs photographed with the IMED-4 device in position
15. Severe co-morbidity or poor general physical/mental health that, in the opinion of the Investigator, will not allow the subject to be a good study candidate (i.e. other disease processes, mental capacity, substance abuse, incarceration, shortened life expectance, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are admitted for inpatient management with acute heart failure syndrome with pulmonary congestion are possible candidates for the study and shall be screened for suitability based on the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2014-07; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Lung Fluid Status | Up to 1 year
  IMED 4 is a new device to measure lung fluid status by assessing how wet or dry the lungs are

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Mass General Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Ohio State University, Columbus, Ohio